CLINICAL TRIAL: NCT04190368
Title: Team Clinic: Virtual Expansion of an Innovative Multi-Disciplinary Care Model for Middle School and High School Adolescents and Young Adults With Type 1 Diabetes
Brief Title: Team Clinic: Virtual Expansion of an Innovative Multi-Disciplinary Care Model for Adolescents and Young Adults With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: University of Southern California (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, jennifer raymond, MD, MCR, Associate Professor of Clinical Pediatrics, Clinical Director of Diabetes Center for Endocrinology, Diabetes, and Metabolism, Vice Chair of the Executive Telehealth Committee, Children's Hospital Los Angeles
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CHLA-19-00062
Record Dates: First submitted 2019-07-22; First posted 2019-12-09 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes
Keywords: Adolescents; Young Adults; Group Medical Visits
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Team Clinic Care: No VTC Groups (Other): Participants attend quarterly visits (1 visit every 3months). Appointments scheduled for Telehealth (TH) (1 in-person visits) as decided by provider/patient and yearly team visit as needed
  • Providers will utilize a patient centered care approach to conducting appointments
  Interventions: Other: Team Clinic Care
- Team Clinic: Virtual Team Clinic Group (Other): Participants will be invited to participate in online/virtual thematic group sessions led by Team Clinic group facilitators (e.g., RD, SW, RN) aimed at improving glycemic control and treatment adherence, increasing social supports and diabetes care satisfaction, and aid in the transition from caregiver led treatment to self care.
  o Patients and Family members attend their own online sessions: Energy Training, Proficiency Training, Resilience Training, Balance Training, Miscellaneous sessions - scheduled as needed
  Interventions: Other: Team Clinic Care
- Standard Care: No VTC Groups (Other): Appointments will continue as usually with provider (quarterly visits; 1 visit every 3 months), but will be referred for necessary care per usual methods (e.g., diabetes education or supportive services).
  Interventions: Other: Standard Care
- Standard Care: Virtual Team Clinic (Other): Appointments will continue as usually with provider (quarterly visits; 1 visit every 3 months), but will be referred for necessary care per usual methods (e.g., diabetes education or supportive services).
  o Patients and Family members attend their own online sessions: Energy Training, Proficiency Training, Resilience Training, Balance Training, Miscellaneous sessions - scheduled as needed
  Interventions: Other: Standard Care

INTERVENTIONS:
Other: Team Clinic Care — Participants attend quarterly visits (1 visit every 3months). Appointments scheduled for Telehealth (TH) (1 in-person visits) as decided by provider/patient.
  Selected providers will be trained in the Team Clinic Care protocol for completing medical appointments. Team Clinic Care key components:
  (1) Shared decision making: Providers, AYA, parent/caregiver will mutually agree on priorities for each medical visit using a shared decision making tool (2) Autonomy supportive care: Providers will be trained in skills building, patient centered key elements, intervention bites, reviewing plans, designed to support AYA autonomy and intrinsic motivation. AYA will also direct extent of eligible family involvement. (3) Goal setting and action planning: Providers will be trained to coach AYA in setting SMART goals, developing action plans, and establishing a plan for follow-up between visits as appropriate. (4) Fidelity Review and process for self-assessment
  Arms: Team Clinic Care: No VTC Groups; Team Clinic: Virtual Team Clinic Group
Other: Standard Care — Participants attend quarterly visits (1 visit every 3 months) and see their diabetes care provider. They do not participate in Team Clinic group visits but if they need diabetes education or supportive services they will be referred for necessary care per usual methods.
  Arms: Standard Care: No VTC Groups; Standard Care: Virtual Team Clinic

SUMMARY:
Team Clinic is a new care approach for middle and high school aged patients living with T1D and their families. This study is a 15-month randomized control trial (RCT) that consists of Virtual Team Clinic Care appointments (primarily telemedicine, and in-person as necessary) and Virtual Team Clinic group appointments with a multidisciplinary diabetes care team. Assignment into 1 of 4 intervention groups Team Clinic Care vs. Standard Care which consist of either Virtual Team Clinic Group or no group.

Groups:

1. Standard Care - No Group
2. Standard Care - Virtual Team Clinic Group
3. Team Clinic Care - No Group
4. Team Clinic Care - Virtual Team Clinic Group Virtual Team Clinic group sessions will be facilitated by clinical care team (e.g., Registered Dietician, Social Worker, Registered Nurse, etc.)

   * Patients and parents will attend their own online session

DETAILED DESCRIPTION:
Team Clinic is an innovative approach to addressing patient developmental, psycho-social, and familial challenges; while also tackling the medical infrastructure and multi-disciplinary care challenges encountered by middle school and high school aged individuals with Type 1 Diabetes and their caregivers. This new approach consists of Team Clinic Care appointments (primarily telemedicine, and in-person as necessary). The study incorporates Virtual Team Clinic group/medical group appointments with a multidisciplinary diabetes care team of diabetes care providers. Each group will have a special theme (thematic group visits) and learning experience aimed at improving glycemic control and treatment adherence, increasing social supports and diabetes care satisfaction, and aid in the transition from caregiver led treatment to self care. Part of the goal of VTC is to spend less time in clinic while still receiving important diabetes education, support, and medical care.

ELIGIBILITY:
Inclusion

1. Diagnosis of type 1 diabetes > 6 month duration
2. Grades 6th, 7th, and 8th ,9th, 10th, 11th, 12th at time of intervention
3. Not currently participating in other group interventions
4. English speaking

Exclusions

1. Severe behavioral or developmental disabilities in parent or child
2. Severe psychological diagnoses in parent or child that would make group participation difficult
3. Significant comorbid medical conditions that would make the patient non-eligible for group participation (e.g. cystic fibrosis, uncontrolled thyroid disease)
4. Non-English speaking

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 79 (Actual)
Dates: Start 2021-09-07 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C at Baseline | baseline to 12 months
  Lab Results: Electronic Medical Record Hemoglobin A1c (HbA1c) %
Hemoglobin A1C Progression | At baseline (0), 3 months, 6 months, 9 months, 12 months
  HbA1c % At-Home Kit
Number of Team Clinic Care cohort participants attending appointments | 12 months
  Attendance will be recorded for each Team Clinic visit
Number of Virtual Team Clinic Care cohort participants completing appointments | 12 months
  Attendance will be recorded for each Virtual Team Clinic Visit
Number of Team Clinic Care cohort participants completing appointments | 12 months
  Electronic Medical Record (EMR) Abstraction
Patient and Provider/Clinic Staff Satisfaction as assessed using the Health Care Climate questionnaire | 12 months
  Likert scale "Very dissatisfied" is 1, "Dissatisfied" is 2, "Neutral" is 3, "Satisfied" is 4, and "Very Satisfied" is 5. Higher scores indicate more satisfaction, lower scores indicate low satisfaction
Patient and Provider/Staff Satisfaction | 12 months
  Cultural Competence Consumer Assessment of Healthcare Providers and Systems (CAHPS) - likert Scale; range 0-10, low range indicates low trust and high values indicate trust.
Patient Experience | 12 months
  Patient Experience Measures Consumer Assessment of Healthcare Providers and Systems (CAHPS) - likert Scale; range 0-10; lower range represents low rating, higher ranges indicate higher rating
Social Determinants of Health Tool | At 0 (baseline)
  Social determinants of health as assessed using a social and environmental factors questionnaire. Polar; Yes or No questions about food insecurity and transportation, "did you worry that your food would run out before you got money to buy more?" "have you or your family ever been unable to go to the doctor because of distance or transportation?"
Number of Standard Clinic cohort participants completing appointments | 12 months
  Attendance will be recorded for each standard care visit
Number of Standard Care cohort participants completing appointments | 12 months
  Electronic Medical Record (EMR) Abstraction

SECONDARY OUTCOMES:
Number of Team Clinic Care cohort participants with diabetic ketoacidosis | 12 months
  Diabetic ketoacidosis events both by self report (i.e., did you have any episodes of diabetic ketoacidosis in the past 3 months) and EMR
Number of Standard Care cohort participants with diabetic ketoacidosis | 12 months
  Diabetic ketoacidosis events both by self report (i.e., did you have any episodes of diabetic ketoacidosis in the past 3 months) and EMR
Number of Team Clinic cohort participants with severe hypoglycemia | 12 months
  Severe hypoglycemia events both by self report (i.e., did you have any episodes of severe hypoglycemia in the past 3 months) and EMR
Number of Standard Care cohort participants with severe hypoglycemia | 12 months
  Severe hypoglycemia events both by self report (i.e., did you have any episodes of severe hypoglycemia in the past 3 months) and EMR
Diabetes Family Conflict Scale | At 0 (baseline) and 12 months (after visit 4)
  Diabetes Family Conflict as assessed using the Diabetes Family Conflict Scale (DFCS) for parents and the DFCS for children. Each scale is a 20 item questionnaire using a Likert Scale (1 = Almost Never, 2 = Sometimes, 3 = Almost Always). Parent and Child questionnaires are combined with a possible score range from 40 to 120 with higher scores indicating more conflict.
Problem Areas in Diabetes in Caregivers | At 0 (baseline) and 12 months (after visit 4)
  Problem Areas in Diabetes as assessed using the Problem Areas in Diabetes - Caregivers (PAID-T). This instrument was designed to assess emotional distress related to caring for a teen with diabetes. It is a 26 item questionnaire using a 6 point Likert Scale format (1-2 = Not a problem, 3-4 = Moderate Problem, 5-6 = Serious Problem). The possible score range is from 26 to 156 with higher scores indicating increased distress.
Problem Areas in Diabetes in Teens | At 0 (baseline) and 12 months (after visit 4)
  Problem Areas in Diabetes as assessed using the Problem Areas in Diabetes - Teens (PAID-T). This instrument was designed to assess emotional distress in teens with diabetes. It is a 26 item questionnaire using a 6 point Likert Scale format (1-2 = Not a problem, 3-4 = Moderate Problem, 5-6 = Serious Problem). The possible score range is from 26 to 156 with higher scores indicating increased distress.
Patient - Practitioner Orientation Scale | At 0 (baseline) and 12 months (after visit 4)
  Patient - Practitioner Orientation Scale consists of 18 items and 2 subscales. It assesses provider beliefs on patient centeredness. 6-point Likert scale: "Strongly disagree," "Moderately Disagree," "Slightly Disagree," "Slightly Agree," "Moderately Agree," and "Strongly Agree." PPOs score is computed by taking the mean of the 18 items with a minimum score being "1" and maximum being "6." Higher scores present more patient-centered attitudes.
Cost to Instituition | 12 months
  Cost to Institution as assessed by Patient Health Utilization questionnaire. Polar; Yes or No questions about health service usage in the last three months, "have you had to be admitted to the hospital?" Open-ended question about number of time health services were used, "how many times were you admitted to the hospital for reasons related to diabetes?"
Cost to Institution - Standard care | 12 months
  Cost to Institution as assessed using the In Person questionnaire. Polar; Yes or No questionnaire about appointment attendance; "did you attend an in-person, standard care appointment?" "How long was your in-person appointment?" Open-ended questions about time, "how long did it take?"
Cost to Institution - Team Clinic | 12 months
  Cost to Institution as assessed using the Online Appointment questionnaire. Polar; Yes or No questions about attendance to in person, Team Clinic care appointment. "Did you attend your in person appointment?" "What types of providers did you see?" Open-ended questions asking about time, "how long did it take?"
Cost to Institution - Clinic Costs | 12 months
  Cost to Institution as assessed using the Clinic Cost, Preparation, and Delivery for Providers and Staff questionnaire. Multiple choice questions about person (Doctor, Nurse and Social Worker) and appointment type provided to patient.
Cost to Institution - Team Costs | 12 months
  Cost to Institution as assessed using Team Costs of Provider and Staff Training questionnaire. Multiple choice questions used to identify person being trained (e.g. role), "Doctor," "Nurse Practitioner," "Social Worker." Polar; Yes or No questions about provider and staff training for Team Clinic appointment; training on, "roles of the attendees," in Team Clinic. Issues regarding the study and study toolkit.
Cost to Institution | 12 months
  Cost to Institution as assessed using the Feasibility and Usability of Toolkit questionnaire. Multiple choice questions used to identify the training session, role, provider, usability of toolkit, and training time. The questionnaire also includes a 6-point Likert scale: "Strongly disagree," "Somewhat Disagree," "Neutral," "Slightly Agree," "Somewhat Agree," and "Strongly Agree."
Clinical Efficiency | 12 months
  Assessed using the Clinical Efficiency questionnaire which captures the number of patients seen during a given time period), team members seen, and time patients spent with team members.
Diabetes Strengths and Resilience Measure for Children | At 0 (baseline) and 12 months (after visit 4)
  DSTAR-Child assesses adaptive aspects of adolescents' diabetes management (i.e., "strengths"), and is related to clinical outcomes. It is a 12 item questionnaire using a 5 point Likert Scale format (1= Never, 2= Rarely, 3= Sometimes, 4= Often, 5= Almost Always). Items are scored on a scale of 12-60.
Diabetes Strengths and Resilience Measure for Teens | At 0 (baseline) and 12 months (after visit 4)
  DSTAR-Teen assesses adaptive aspects of adolescents' diabetes management (i.e., "strengths"), and is related to clinical outcomes. It is a 12 item questionnaire using a 5 point Likert Scale format (1= Never, 2= Rarely, 3= Sometimes, 4= Often, 5= Almost Always). Items are scored on a scale of 12-60.
PROMIS - Peds Peer Relationships | At 0 (baseline) and 12 months (after visit 4)
  Patient-Reported Outcomes Measurement Information System (PROMIS )- Peds Peer Relationships. Evaluates and monitors social health. Likert scale used to assess quality of relationships with friends and acquaintances. (1= Never, 2= Almost Never, 3= Sometimes, 4=Often, 5= Almost Always)
PROMIS - Peds Family Relationships | At 0 (baseline) and 12 months (after visit 4)
  Patient-Reported Outcomes Measurement Information System (PROMIS )- Peds Family Relationships. Evaluates and monitors social health. Likert scale used to assess the subjective (affective, emotional, cognitive) experience of being involved with one's family, feeling like an important person in the family, of feeling accepted and cared for, and feeling that family members, especially parents, can be trusted and depended on for help and understanding. (1= Never, 2= Almost Never, 3= Sometimes, 4=Often, 5= Almost Always)
PROMIS - Emotional Support | At 0 (baseline) and 12 months (after visit 4)
  Patient-Reported Outcomes Measurement Information System (PROMIS )- Emotional Support (Parents/caregivers). Evaluates and monitors social health. Likert scale assessing perceived feelings of being cared for and valued as a person; having confidant relationships. (1= Never, 2= Almost Never, 3= Sometimes, 4=Often, 5= Almost Always)
PROMIS - Instrumental Support | At 0 (baseline) and 12 months (after visit 4)
  Patient-Reported Outcomes Measurement Information System (PROMIS )- Instrumental Support (Parents/caregivers). Evaluates and monitors social health. Likert scale assessing Perceived availability of assistance with material, cognitive or task performance. (1= Never, 2= Almost Never, 3= Sometimes, 4=Often, 5= Almost Always)
PROMIS - Informational Support | At 0 (baseline) and 12 months (after visit 4)
  Patient-Reported Outcomes Measurement Information System (PROMIS )- Informational Support (Parents/caregivers). Evaluates and monitors social health. Likert scale assessing Perceived availability of helpful information or advice.. (1= Never, 2= Almost Never, 3= Sometimes, 4=Often, 5= Almost Always)

OTHER OUTCOMES:
Socio-Demographic History | At 0 (baseline)
  Self-reported demographic history (gender, age, race, household income, etc) will be collected.
Medical History | 12 months
  General health history via self report and EMR
Diabetes Treatment Regimen - glucometer | 12 months
  Diabetes treatment regimen assessed through blood glucose checks per day from glucometer downloads will be collected from devices and EMR.
Diabetes Treatment Regimen - insulin pump | 12 months
  Diabetes treatment regimen assessed through insulin boluses per day from insulin pump downloads will be collected from devices and EMR.
Diabetes Treatment Regimen - continuous glucose monitors | 12 months
  Diabetes treatment regimen assessed through percentage of glucose values low, in target, or high for patients on continuous glucose monitors will be collected from devices and EMR.
Self-care and mobility as assessed using the EuroQOL five dimensions five levels youth (EQ-5D-Y) questionnaire | At 0 (baseline) and 12 months (after visit 4)
  Likert scale; used to measure respondents' endorsement of particular statements. Descriptive system top answer is 1 and last answer is 5. Missing items will be coded as 9. Online software used to score.
The Child Health Utility | At 0 (baseline) and 12 months (after visit 4)
  The Child Health Utility 9 dimensions assesses health-related quality of life (HRQoL). Multiple choice used to capture respondents' endorsement of particular statements about experience. "I don't feel [upset] today," "I feel a little bit [upset] today," "I feel a bit [upset] today," "I feel quite [upset] today," "I feel very [upset] today"
Patient Health Questionnaire-8 (PHQ-8) | At 0 (baseline) and 12 months (after visit 4)
  Composed of 8 items to screen, diagnose, and measure the severity of depression.
Shared Medical Appointments - Patient/AYA | baseline to 12 months
  Likert scale; "Strongly disagree" is 1, "disagree" is 2, "neutral" is 3, "agree" is 4, "strongly agree" is 5. Also, includes 3 open-ended questions to measures satisfaction for shared medical appointments.
Shared Medical Appointments- Parent/caregiver | baseline to 12 months
  Likert scale;"Strongly disagree" is 1, "disagree" is 2, "neutral" is 3, "agree" is 4, "strongly agree" is 5. Also, includes 3 open-ended questions to measures satisfaction for shared medical appointments.
Self Care - Related to Diabetes as assessed by Self-Care questionnaire | baseline to 12 months
  Multiple Choice. Questions about diabetes related self care, "How many hours per day do you currently devote to managing your glucose levels?"
Diabetes Family Responsbility Questionnaire - Parent | At 0 (baseline) and 12 months (after visit 4)
  Asseses how adolescents with T1D and their families/caregivers share diabetes management and responsibilities. 17 item questionnaire with a 3 factor solution. "Child" is 1, "equal" is 2, and "parent" is 3. A higher score indicates higher levels of caregiver/parent/family responsbility for diabetes management.
Diabetes Family Responsbility Questionnaire - Teen | At 0 (baseline) and 12 months (after visit 4)
  Asseses how parents/caregivers of children/teens living with T1D share diabetes management and responsibilities. 17 item questionnaire with a 3 factor solution. "Child" is 1, "equal" is 2, and "parent" is 3. A higher score indicates higher levels of caregiver/parent/family responsbility for diabetes management.
Clinical Variables | At 0 (baseline) and 12 months (after visit 4)
  Polar; Yes or No questionnaire. Data extracted from EMR : cholesterol, high density lipoprotein, triglycerides, smoking status, nephropathy, microalbuminaria, macroalbuminaria, end-stage renal disease (death from end-stage renal disease), neuropathy, peripheral arterial disease (low extremity amputation), retinopathy (proliferative retinopathy), macular edema, blindness, angina, myocardial infarction, stroke, heart failure, revascularization (Coronary artery bypass grafting, PCA, and stenting). If answered "yes" for the following: ergosterol, HDL,microalbuminaria, and macroalbuminaria, values will be recorded.
ADA and CCS standards | 12 months
  EMR abstraction: Questions assess compliance with ADA and CCS standards when patients have contact with all team members annually. This will be noted with polar questions "Yes" or No." This will be tracked for all patients in the study (e.g., Team Clinic and Standard Clinic).
Single Item Literacy Scale | At 0 (Baseline) and 12 months (after visit 4)
  Literacy assessed using the Single Item Literacy Scale. Multiple choice question asking about suppoort needed with reading materials. Options, "never," "rarely," "sometimes," "often," "always"
Provider Centered Care Observation Form (PCOF) | 12 months
  Assessing the fidelity of care delivery for ensuring that patients receive full benefits of the Team Clinic intervetion. Domain checklist, "Establishes Rapport," "Maintain Relationship Throughout the Visit," "Collaborative upfront agenda setting," "Maintain Efficiency using transparent thinking and respectful interruption," "Gathering information," "Assessing patient or family perspective on health," "Electronic Medical Record Use," "Physical Exam"
Facilitator Centered Care Observation Form (PCOF) | 12 months
  Assessing the fidelity of care delivery for ensuring that patients receive full benefits of the Team Clinic intervetion. Domain checklist, "Establishes Rapport," "Maintains Relationship Trhoughout the Visit," "Session Introduction and Icebreaker," "Session Preparation," "Gathering Information," "Assessing Patient or Family Persepctive on Health/Understanding Context," "Blood Glucose Charting," "Blood Glucose Discussion," "Activity Kit Review"
Provider/Facilitator Session Feedback Form: | 12 months
  Assess provider experience during clinic visit and patient-center delivery. Multiple choice, "Establishing Rapport and Maintaining Relationship," "Agenda-setting, Thinking Out-Loud, and Collaboration," "Gathering Information and Understanding Context," "EMR Review and Physical Exam," "Promoting Behavior Change or Self-Management," "Collaborative Planning and Closure," "None of these"

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer K Raymond, MD, MCR, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Development, execution, and data collection for this study is completed with a Principle Investigator at Children's Hospital Los Angeles. With documented permission of the IRB, a PI may develop a de-identified database, codebook, and mechanism by which data can be shared with qualified investigators. Interested Investigators will complete a request form stating the aims of their analyses, analytic plan, available resources for completing a project, timeline, and goals (i.e. manuscripts or grant applications). The PIs and their research team will review requests to determine whether the analyses constitute an innovative exploration of the data, whether the team has resources to complete the request, and whether data will be adequately protected and managed. If issues arise, the PIs and research team will negotiate a fair resolution with interested investigators and NIH staff.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: Data will be available within 6 months of study completion.
Access Criteria: Data access requests will be reviewed, and requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Background] Miller KM, Foster NC, Beck RW, Bergenstal RM, DuBose SN, DiMeglio LA, Maahs DM, Tamborlane WV; T1D Exchange Clinic Network. Current state of type 1 diabetes treatment in the U.S.: updated data from the T1D Exchange clinic registry. Diabetes Care. 2015 Jun;38(6):971-8. doi: 10.2337/dc15-0078. PMID 25998289
- [Background] Reiss J, Gibson R. Health care transition: destinations unknown. Pediatrics. 2002 Dec;110(6 Pt 2):1307-14. PMID 12456950
- [Background] Peters A, Laffel L; American Diabetes Association Transitions Working Group. Diabetes care for emerging adults: recommendations for transition from pediatric to adult diabetes care systems: a position statement of the American Diabetes Association, with representation by the American College of Osteopathic Family Physicians, the American Academy of Pediatrics, the American Association of Clinical Endocrinologists, the American Osteopathic Association, the Centers for Disease Control and Prevention, Children with Diabetes, The Endocrine Society, the International Society for Pediatric and Adolescent Diabetes, Juvenile Diabetes Research Foundation International, the National Diabetes Education Program, and the Pediatric Endocrine Society (formerly Lawson Wilkins Pediatric Endocrine Society). Diabetes Care. 2011 Nov;34(11):2477-85. doi: 10.2337/dc11-1723. No abstract available. PMID 22025785
- [Background] Rosen DS, Blum RW, Britto M, Sawyer SM, Siegel DM; Society for Adolescent Medicine. Transition to adult health care for adolescents and young adults with chronic conditions: position paper of the Society for Adolescent Medicine. J Adolesc Health. 2003 Oct;33(4):309-11. doi: 10.1016/s1054-139x(03)00208-8. No abstract available. PMID 14519573
- [Background] Bryden KS, Dunger DB, Mayou RA, Peveler RC, Neil HA. Poor prognosis of young adults with type 1 diabetes: a longitudinal study. Diabetes Care. 2003 Apr;26(4):1052-7. doi: 10.2337/diacare.26.4.1052. PMID 12663572
- [Background] Sanchez I. Implementation of a diabetes self-management education program in primary care for adults using shared medical appointments. Diabetes Educ. 2011 May-Jun;37(3):381-91. doi: 10.1177/0145721711401667. Epub 2011 Mar 31. PMID 21454887
- [Background] Rising SS. Centering pregnancy. An interdisciplinary model of empowerment. J Nurse Midwifery. 1998 Jan-Feb;43(1):46-54. doi: 10.1016/s0091-2182(97)00117-1. PMID 9489291
- [Background] Noffsinger E. Enhance satisfaction with drop-in group visits. . Hippocrates. 2001;15(2):30-36.
- [Background] Noffsinger EB. Running Group Visits in Your Practice. New York, NY: Springer Science+Business Media; 2009.
- [Background] Floyd BD, Block JM, Buckingham BB, Ly T, Foster N, Wright R, Mueller CL, Hood KK, Shah AC. Stabilization of glycemic control and improved quality of life using a shared medical appointment model in adolescents with type 1 diabetes in suboptimal control. Pediatr Diabetes. 2017 May;18(3):204-212. doi: 10.1111/pedi.12373. Epub 2016 Feb 26. PMID 26919322
- [Background] Raymond JK, Shea JJ, Berget C, Cain C, Fay-Itzkowitz E, Gilmer L, Hoops S, Owen D, Shepard D, Spiegel G, Klingensmith G. A novel approach to adolescents with type 1 diabetes: the team clinic model. Diabetes Spectr. 2015 Jan;28(1):68-71. doi: 10.2337/diaspect.28.1.68. No abstract available. PMID 25717281
- [Background] Hood KK, Butler DA, Anderson BJ, Laffel LM. Updated and revised Diabetes Family Conflict Scale. Diabetes Care. 2007 Jul;30(7):1764-9. doi: 10.2337/dc06-2358. Epub 2007 Mar 19. PMID 17372149
- [Background] Evans M, Davis, L, & Weissberg-Benchell, J. Psychometric properties of the child and parent problem areas in diabetes measures. Paper presented at: Poster presented at the 76th Annual Scientific Sessions of the American Diabetes AssociationJune, 2016; New Orleans, Louisiana.
- [Background] Weissberg-Benchell J, Antisdel-Lomaglio J. Diabetes-specific emotional distress among adolescents: feasibility, reliability, and validity of the problem areas in diabetes-teen version. Pediatr Diabetes. 2011 Jun;12(4 Pt 1):341-4. doi: 10.1111/j.1399-5448.2010.00720.x. Epub 2011 Mar 28. PMID 21443583
- [Background] McClain MR, Klingensmith GJ, Anderson B, Berget C, Cain C, Shea J, Campbell K, Pyle L, Raymond JK. Team Clinic: Group Approach to Care of Early Adolescents With Type 1 Diabetes. Diabetes Spectr. 2018 Aug;31(3):273-278. doi: 10.2337/ds17-0063. No abstract available. PMID 30140144
- [Background] Raymond JK. Models of Care for Adolescents and Young Adults with Type 1 Diabetes in Transition: Shared Medical Appointments and Telemedicine. Pediatr Ann. 2017 May 1;46(5):e193-e197. doi: 10.3928/19382359-20170425-01. PMID 28489225
- [Background] Rijswijk C, Zantinge E, Seesing F, Raats I, van Dulmen S. Shared and individual medical appointments for children and adolescents with type 1 diabetes; differences in topics discussed? Patient Educ Couns. 2010 Jun;79(3):351-5. doi: 10.1016/j.pec.2010.04.016. Epub 2010 May 2. PMID 20439147
- [Background] Noordman J, van Dulmen S. Shared Medical Appointments marginally enhance interaction between patients: an observational study on children and adolescents with type 1 diabetes. Patient Educ Couns. 2013 Sep;92(3):418-25. doi: 10.1016/j.pec.2013.06.008. Epub 2013 Jul 3. PMID 23830238
- [Background] Mejino A, Noordman J, van Dulmen S. Shared medical appointments for children and adolescents with type 1 diabetes: perspectives and experiences of patients, parents, and health care providers. Adolesc Health Med Ther. 2012 Jun 15;3:75-83. doi: 10.2147/AHMT.S32417. eCollection 2012. PMID 24600288
- [Background] Berget C, Lindwall J, Shea JJ, Klingensmith GJ, Anderson BJ, Cain C, Raymond JK. Team Clinic: An Innovative Group Care Model for Youth with Type 1 Diabetes-Engaging Patients and Meeting Educational Needs. J Nurse Pract. 2017 Jun;13(6):e269-e272. doi: 10.1016/j.nurpra.2017.03.016. Epub 2017 Apr 26. PMID 28993721
- [Background] Willi SM, Miller KM, DiMeglio LA, Klingensmith GJ, Simmons JH, Tamborlane WV, Nadeau KJ, Kittelsrud JM, Huckfeldt P, Beck RW, Lipman TH; T1D Exchange Clinic Network. Racial-ethnic disparities in management and outcomes among children with type 1 diabetes. Pediatrics. 2015 Mar;135(3):424-34. doi: 10.1542/peds.2014-1774. PMID 25687140
- [Background] Hays RD, Shaul JA, Williams VS, Lubalin JS, Harris-Kojetin LD, Sweeny SF, Cleary PD. Psychometric properties of the CAHPS 1.0 survey measures. Consumer Assessment of Health Plans Study. Med Care. 1999 Mar;37(3 Suppl):MS22-31. doi: 10.1097/00005650-199903001-00003. PMID 10098556
- [Background] Morris NS, MacLean CD, Chew LD, Littenberg B. The Single Item Literacy Screener: evaluation of a brief instrument to identify limited reading ability. BMC Fam Pract. 2006 Mar 24;7:21. doi: 10.1186/1471-2296-7-21. PMID 16563164
- [Background] Whittemore R, Jaser S, Chao A, Jang M, Grey M. Psychological experience of parents of children with type 1 diabetes: a systematic mixed-studies review. Diabetes Educ. 2012 Jul-Aug;38(4):562-79. doi: 10.1177/0145721712445216. Epub 2012 May 11. PMID 22581804
- [Background] Continous Glucose Monitoring (CGM) as a CCS/GHPP Program Benefit [press release]. 3/6/2017.
- [Background] American Diabetes Association. Erratum. Glycemic Targets. Sec. 6. In Standards of Medical Care in Diabetes-2017. Diabetes Care 2017;40(Suppl. 1);S48-S56. Diabetes Care. 2017 Jul;40(7):985. doi: 10.2337/dc17-er07a. Epub 2017 May 18. No abstract available. PMID 28522557
- [Background] Winkley K, Ismail K, Landau S, Eisler I. Psychological interventions to improve glycaemic control in patients with type 1 diabetes: systematic review and meta-analysis of randomised controlled trials. BMJ. 2006 Jul 8;333(7558):65. doi: 10.1136/bmj.38874.652569.55. Epub 2006 Jun 27. PMID 16803942
- [Background] Kahana S, Drotar D, Frazier T. Meta-analysis of psychological interventions to promote adherence to treatment in pediatric chronic health conditions. J Pediatr Psychol. 2008 Jul;33(6):590-611. doi: 10.1093/jpepsy/jsm128. Epub 2008 Jan 11. PMID 18192300
- [Background] Hilliard ME, Harris MA, Weissberg-Benchell J. Diabetes resilience: a model of risk and protection in type 1 diabetes. Curr Diab Rep. 2012 Dec;12(6):739-48. doi: 10.1007/s11892-012-0314-3. PMID 22956459
- [Background] Rubin RY-H, D; Peyrot, M. Parent-child responsibility and conflict in diabetes care (Abstract) Diabetes Care. 1989;38:28A.
- [Background] Palladino DK, Helgeson VS. Friends or foes? A review of peer influence on self-care and glycemic control in adolescents with type 1 diabetes. J Pediatr Psychol. 2012 Jun;37(5):591-603. doi: 10.1093/jpepsy/jss009. Epub 2012 Mar 29. PMID 22460759
- [Background] Chiang JL, Kirkman MS, Laffel LM, Peters AL; Type 1 Diabetes Sourcebook Authors. Type 1 diabetes through the life span: a position statement of the American Diabetes Association. Diabetes Care. 2014 Jul;37(7):2034-54. doi: 10.2337/dc14-1140. No abstract available. PMID 24935775
- [Derived] Salvy SJ, Ruelas V, Majidi S, Thomas A, Ashwal G, Reid M, Fox DS, McClain S, Raymond JK. Team clinic: Expansion of a multidisciplinary care model for adolescents with type 1 diabetes. Contemp Clin Trials. 2020 Aug;95:106079. doi: 10.1016/j.cct.2020.106079. Epub 2020 Jul 4. PMID 32634486